CLINICAL TRIAL: NCT01255189
Title: Measurement of the Effect of Positional Changes on Cerebral Oxygenation in Preterm Infants: A Near Infrared Spectroscopy Study
Brief Title: Measurement of the Effect of Positional Changes on Cerebral Oxygenation in Preterm Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Gamze Demirel, Neonatal Intensive Care Unit ( Zekai Tahir Burak Maternity and Teaching Hospital )
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3498
Record Dates: First submitted 2010-12-02; First posted 2010-12-07 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2010-12

CONDITIONS: pOSitional Changes of Premature Infants
Keywords: NIRS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device: near infrared spectroscopy: invos 5100 (Experimental): NIRS device used in this study, the optical field includes a volume of tissue approximately 2 cm deep to the surface probe with a 4-mm source-detector distance, and thus, organ-specific monitoring is feasible in small patients. With informed consent, we applied NIRS probes to the forehead and the lower extremity for cerebral (rSO2C) and peripheric (rSO2P) regional oxygen saturation measurements
  Interventions: Device: Device: near infrared spectroscopy: INVOS 5100; Device: invos 5100

INTERVENTIONS:
Device: Device: near infrared spectroscopy: INVOS 5100 — NIRS device used in this study, the optical field includes a volume of tissue approximately 2 cm deep to the surface probe with a 4-mm source-detector distance, and thus, organ-specific monitoring is feasible in small patients. With informed consent, we applied NIRS probes to the forehead and the lower extremity for cerebral (rSO2C) and peripheric (rSO2P) regional oxygen saturation measurements.
  Other Names: invos 5100
Device: invos 5100 — near infrared spectroscopy: invos 5100

SUMMARY:
Near infrared spectroscopy offers the possibility of noninvasive and continuous bedside investigation of cerebral oxygenation in newborn infants. Using this technique we investigated the effect of positional changes on cerebral oxygenation in preterm infants.

DETAILED DESCRIPTION:
The changes in cerebral perfusion have an important role on the development of intraventricular hemorrhage and periventricular leucomalacia. Near infrared spectroscopy offers the possibility of noninvasive and continuous bedside investigation of cerebral oxygenation in newborn infants. Using this technique we investigated the effect of positional changes on cerebral oxygenation in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

1. <32 gestational age and/or <1500gr.
2. >30th day preterm infants

Exclusion Criteria:

1. sepsis
2. shock
3. severe intracranial hemorrhage
4. NEC
5. abdominal and cranial surgery

Ages: 3 Days to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The effect of positional changes on cerebral oxygenation in preterm infants | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Demirel, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Demirel G, Oguz SS, Celik IH, Erdeve O, Dilmen U. Cerebral and mesenteric tissue oxygenation by positional changes in very low birth weight premature infants. Early Hum Dev. 2012 Jun;88(6):409-11. doi: 10.1016/j.earlhumdev.2011.10.005. Epub 2011 Nov 15. PMID 22088784